CLINICAL TRIAL: NCT04484519
Title: Recovery of Biographical Memories Associated With a Melody: a Functional Magnetic Resonance Imaging Study
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MEMORIA&MUSICA/BBRC2019
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitively unimpaired
  Interventions: Other: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging — Functional Magnetic Resonance Imaging

SUMMARY:
This study aims to validate a functional MRI paradigm to determine the regions involved in the retrieve of music-linked memories

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women (aged 20 - 50)
* Signature of the study's informed consent form, accepting to not receive information with regards to any research results that are not clinically relevant.
* Persons that accept the study's procedure: magnetic resonance imaging.

Exclusion Criteria:

* Contraindication to MRI scanning or conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
* Persons with severe or profound hearing loss or deafness

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Cognitively unimpaied, 20-50 years old
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
fMRI paradigm | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- BarcelonaBeta Brain Research Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided